CLINICAL TRIAL: NCT00770003
Title: A Double-blind, Placebo Controlled, Randomized, Parallel Group Study to Investigate the Tolerability, Safety, Pharmacodynamics and Pharmacokinetics of Repeated Weekly Doses of AZD8848 Administered Intranasally to Seasonal Allergic Rhinitis Patients
Brief Title: Tolerability/PoP Study in Allergic Rhinitis After Intranasal Administration of AZD8848
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0540C00003
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Rhinitis
Keywords: patients; allergic rhinitis; tolerability; safety; nasal symptoms
MeSH Terms: conditions — Rhinitis, Allergic | interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8848
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8848 — nasal spray solution; 30 or 60 µg administered intranasally once weekly for one month
  Arms: 1
Drug: Placebo — nasal spray solution. Once weekly intranasal administrations for one month.
  Arms: 2

SUMMARY:
The primary purpose is to investigate tolerability/safety of repeated weekly doses of AZD8848 administered intranasally to seasonal allergic rhinitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of birch and/ or timothy grass pollen induced seasonal allergic rhinitis for at least the previous 2 years (verified by a positive skin prick test)
* Patients with need of treatment for their nasal symptoms during the pollen season

Exclusion Criteria:

* Clinical relevant disease or abnormality (past or present) - other than allergic rhinitis
* Symptomatic perennial allergic or non-allergic rhinitis
* A history of asthma

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Incidence/nature of adverse events,pulse, BP, body temperature, ECG parameters, lab assessments | During the study
Nasal symptoms, peak nasal inspiratory flow | During the study

SECONDARY OUTCOMES:
Reflective Total Nasal Symptom Score, Peak Nasal Inspiratory Flow | During the study
Blood biomarkers and nasal lavage biomarkers | During the study
Pharmacokinetics | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Greiff, MD PhD, Principal Investigator — Lund University Hospital; Leif T Eriksson, MD, PhD, Study Director — AstraZeneca
Locations (2):
- Sweden (2):
  - Research Site, Helsingborg
  - Research Site, Lund

REFERENCES:
- [Derived] Greiff L, Ahlstrom-Emanuelsson C, Alenas M, Almqvist G, Andersson M, Cervin A, Dolata J, Lindgren S, Martensson A, Young B, Widegren H. Biological effects and clinical efficacy of a topical Toll-like receptor 7 agonist in seasonal allergic rhinitis: a parallel group controlled phase IIa study. Inflamm Res. 2015 Nov;64(11):903-15. doi: 10.1007/s00011-015-0873-2. Epub 2015 Sep 5. PMID 26342289
- [Derived] Greiff L, Cervin A, Ahlstrom-Emanuelsson C, Almqvist G, Andersson M, Dolata J, Eriksson L, Hogestatt E, Kallen A, Norlen P, Sjolin IL, Widegren H. Repeated intranasal TLR7 stimulation reduces allergen responsiveness in allergic rhinitis. Respir Res. 2012 Jun 22;13(1):53. doi: 10.1186/1465-9921-13-53. PMID 22726593
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1657&filename=D0540C00003_Study_Synopsis.pdf